CLINICAL TRIAL: NCT01249729
Title: 3D Reconstructed Image Processin by Computer Proram
Brief Title: 3D Reconstructed Image Processin by Computer Proram From MRI Data
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Taipei Medical University-Wan Fang Hospital, Institutional Review Board
Other Study IDs: 97015
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2008-08

CONDITIONS: 3D Reconstructed Image by Software.
Keywords: Magnetic Resonance Imaging, 3D reconstructed image

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We use the three-dimensional image software reconstruct MRI. The propose of this research purposes as follows: 1. 3D reconstructed image processing from MRI to realize the short term nervous system response after dynamic acupuncture stimulation.2. Realizing the corresponding area in the brain caused by electroacupuncture. 3. Realizing the connection between electroacupuncture stimulation and brain physics, chemistry, and physiology. The implement the two-dimentional image into three-dimensional image by Amira software, in order to find out the difference of the pre-and post- response of the nervous system. In addition, we will use "describe statistics" and "Paired t-test" statistical analysis, compare the statistical difference of blood oxygen concentration.

DETAILED DESCRIPTION:
We use the three-dimensional image software reconstruct MRI. The propose of this research purposes as follows: 1. 3D reconstructed image processing from MRI to realize the short term nervous system response after dynamic acupuncture stimulation.2. Realizing the corresponding area in the brain caused by electroacupuncture. 3. Realizing the connection between electroacupuncture stimulation and brain physics, chemistry, and physiology. The implement the two-dimentional image into three-dimensional image by Amira software, in order to find out the difference of the pre-and post- response of the nervous system. In addition, we will use "describe statistics" and "Paired t-test" statistical analysis, compare the statistical difference of blood oxygen concentration.

Anticipate of results: Using the three-dimensional software reconstruct magnetic resonance imaging to realize the immediate response of nervous system after acupoint acupuncture stimulation, and find out the meridian, nerve or physiological corresponding relationship. It will be a tremendous finding to the world if we can deliver a brain mapping concerning the localization of the response on the central nervous system after various acupoints stimulation.

ELIGIBILITY:
Inclusion Criteria:

* The outpatient service or the in-patient, diagnoses after pediatric nerve doctor, must carry on the central nervous system MRI.

Exclusion Criteria:

* Not symbol cooperation brain MRI condition

Ages: 1 Year to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study expect to seek 100 patients to use the magnetic resonance imaging of brain before and after the acupoint electroacupuncture, measuring the response of all the brain activities, and then implement the two-dimentional image into three-dimensional image by Amira software.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Study Completion 2009-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ein-Yiao Shen, MD, Study Chair — Taipei Medical University-Wan Fong Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan